CLINICAL TRIAL: NCT06535438
Title: The Role of Noncontrast Computed Tomography Markers in Predicting the Clinical Outcome of Cerebral Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Jin Hu (Other)
Responsible Party: Sponsor-Investigator, Jin Hu, Huashan Hospital, Fudan University, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: FDHS2024
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: ICH
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The prognosis of cerebral hemorrhage is good at 90 days
- The prognosis of cerebral hemorrhage is poor at 90 days

SUMMARY:
The goal of this observational study is to To investigate the ability of Noncontrast Computed Tomography to predict clinical prognosis in Intracerebral Hemorrhage.

The main question it aims to answer is:How to judge the prognosis of patients with cerebral hemorrhage by CT image reading at admission.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. had completed a CT examination within 24 h of disease onset;
3. had a hemorrhage that was located in the brain parenchyma, including the basal ganglia, thalamus,brain lobes, brainstem, and cerebellum.

Exclusion Criteria:

1. had secondary ICH caused by brain trauma,cerebrovascular malformations, aneurysms, and tumors;
2. had ischemic cerebral infarction hemorrhagic transformation;
3. had undergone surgical treatment (e.g.hematoma removal or puncture drainage) before the CT examination;
4. had images of poor quality that could notbe accurately evaluated;
5. had a hematoma withborders that could not be delineated, thus precluding delineation of the region of interest (ROI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cerebral hemorrhage who met the criteria and were admitted continuously within the time period
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The prognosis of cerebral hemorrhage at 90 days | 90 days
  The Modified Rankin Scale was used to evaluate the prognosis of the patients, and MRS Score >2 indicated poor prognosis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei L, Wu B, Guo T, Ru D, Gao C, Wu J, Wu A, Yue H, Hu J, Wei L, Geng Z, Wang K. Development and validation of a machine learning-based model for 90-day prognosis outcome in spontaneous intracerebral hemorrhage patients based on non-contrast computed tomography: a multicenter retrospective observational study. EClinicalMedicine. 2025 Sep 12;88:103507. doi: 10.1016/j.eclinm.2025.103507. eCollection 2025 Oct. PMID 41181845